CLINICAL TRIAL: NCT00916656
Title: Efficacy and Safety of Fibrinogen Concentrate (Human) (FCH) for On-demand Treatment of Acute Bleeding in Subjects With Congenital Fibrinogen Deficiency
Brief Title: Fibrinogen Concentrate (Human) - Efficacy and Safety Study
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BI3023_3001; 1475 (Other: CSL Behring); 2007-004088-22 (EudraCT Number)
Record Dates: First submitted 2009-06-08; First posted 2009-06-09 (Estimated); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Afibrinogenemia; Hypofibrinogenemia; Fibrinogen Deficiency
Keywords: Congenital fibrinogen deficiency
MeSH Terms: conditions — Afibrinogenemia | interventions — Fibrinogen; cryoprecipitate coagulum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prospective Arm (Experimental)
  Interventions: Biological: Fibrinogen Concentrate, Human (FCH)
- Historical Control (Other)
  Interventions: Biological: Cryoprecipitate

INTERVENTIONS:
Biological: Fibrinogen Concentrate, Human (FCH) — Intravenous (IV) infusion to reach the peak target levels of 100 mg/dL with an accepted lower limit of 80 mg/dL on at least 3 subsequent days for minor bleeding episodes and 150 mg/dL with an accepted lower limit of 130 mg/dL on at least 7 subsequent days for major bleeding episodes.
  If a subject's fibrinogen level is not known on Day 1, at the time treatment is initiated for the acute bleed (e.g., because they did not have a screening visit), the starting dose is to be 70 mg/kg b.w. Otherwise, the dose will be calculated individually.
  Other Names: Haemocomplettan P; RIASTAP
  Arms: Prospective Arm
Biological: Cryoprecipitate — Patients that received on-demand treatment with Cryoprecipitate for a classified bleeding event (minor or major) with a documented hemostatic efficacy assessment.
  Arms: Historical Control

SUMMARY:
This is a multinational, multicenter, prospective, open-label historically controlled Phase IIIb non-inferiority clinical trial on the efficacy and safety of Fibrinogen Concentrate (Human).

It is estimated that 150-300 patients in the U.S. suffer from afibrinogenemia. Substitution with cryoprecipitate or alternative treatments have limited safety and efficacy.

The primary purpose of the study is to demonstrate the hemostatic efficacy of Fibrinogen Concentrate (Human) by adequately controlling acute bleeding (spontaneous or after trauma) in patients with congenital fibrinogen deficiency (afibrinogenemia and hypofibrinogenemia). Cryoprecipitate hemostatic efficacy data from a retrospective physician survey will be used as a historical control.

ELIGIBILITY:
Inclusion Criteria:

* Documented congenital fibrinogen deficiency (afibrinogenemia and hypofibrinogenemia), expected to require treatment for bleeding
* Presenting with an episode of acute bleeding (either spontaneous or after trauma) not requiring surgery
* Provide informed consent

Exclusion Criteria:

* Life expectancy < 6 months
* Bleeding disorder other than congenital fibrinogen deficiency, but including dysfibrinogenemia
* Treatment with any investigational medicinal product (IMP) in the 30 days prior to enrollment
* Treatment with any fibrinogen concentrate or other fibrinogen containing blood product in the 2 weeks prior to enrollment
* Treatment with any coagulation active drug (i.e., non-steroidal-antirheumatics, warfarin, cumarin derivates, platelet aggregation inhibitors) in 1 week prior to enrollment or as a planned or expected medication during the time period from Day 1 until 24 hours after the last FCH infusion
* Presence or history of hypersensitivity to FCH
* Presence or history of deep vein thrombosis or pulmonary embolism within 1 year prior to enrollment
* Presence or history of arterial thrombosis within 1 year prior to enrollment
* Presence or history of hypersensitivity to human plasma proteins
* Presence or history of esophageal varicose bleeding
* End stage liver disease (i.e., Child Pugh score B or C)
* Planned or expected surgery (i.e., for bleedings from aneurysm or splenic rupture)
* Pregnancy, or an intention to become pregnant during the study
* Currently breast-feeding, or with the intention of breast-feeding during the study
* Human immunodeficiency virus (HIV) positive
* Polytrauma, present or within 6 months prior to enrollment
* Suspicion of an anti-fibrinogen inhibitor as indicated by previous in-vivo recovery (IVR), if available (< 0.5 (mg/dL)/(mg/kg))
* Previous inclusion and treatment in the prospective part of the study
* Participation in any clinical study in the 30 days prior to enrollment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-10; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Clinical assessment of hemostatic efficacy | 24 hours after last infusion or at Day 14 (whichever occurs first)

SECONDARY OUTCOMES:
Maximum clot firmness (MCF) | Prior to and 60 minutes after the end of each infusion
Fibrinogen plasma level | 60 minutes, 3 hours, 6 hours, and 12 hours after the end of the first infusion; before and 60 minutes after each subsequent infusion
In vivo recovery of fibrinogen | 60 minutes, 3 hours, 6 hours and 12 hours after the end of the first infusion; before and 60 minutes after the end of each subsequent infusion and at the time of the overall clinical assessment of hemostatic efficacy
Virus safety markers | Day 1 to Day 45

CONTACTS AND LOCATIONS:
Overall Officials: Program Director, Clinical R&D, Study Director — CSL Behring